CLINICAL TRIAL: NCT00221962
Title: The Cognitive Effects of Aripiprazole in Children
Brief Title: Study of Aripiprazole (Abilify) in Children With ADHD (Attention Deficit Hyperactivity Disorder)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospitals Cleveland Medical Center (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Principal Investigator, Robert L Findling, MD, Director, Child and Adolescent Psychiatry, University Hospitals Cleveland Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: cognition
Record Dates: First submitted 2005-09-16; First posted 2005-09-22 (Estimated); Last update posted 2014-12-15 (Estimated); Status verified 2013-06

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Aripiprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Open label treatment with aripiprazole (Other): After 1-3 week screening phase, entered six week open trial of aripiprazole initiated at 2.5mg/day. DOsing was increased weekly in 2.5mg increments in order to reach maximum dose of 10mg/d.
  Interventions: Drug: Aripiprazole

INTERVENTIONS:
Drug: Aripiprazole — Open label
  Other Names: As previously described.

SUMMARY:
To look at the cognitive effects of abilify in children with a primary diagnosis of Attention Deficit Hyperactivity Disorder. To examine the safety, effectiveness and tolerability of abilify in children with a primary diagnosis of Attention Deficit Hyperactivity Disorder.

DETAILED DESCRIPTION:
This will be a prospective, open-label, 6-week trial of APZ in outpatient children 8-12 years of age with a primary diagnosis of ADHD free of other major psychopathology. The six-week treatment phase will be proceeded by a 1-3 week screening phase.

The study cohort will consist of 10 children with ADHD combined type and 10 children with ADHD predominantly inattentive type who complete the study.

Cognitive measures will be assessed prior to APZ therapy and after 6 weeks of APZ treatment.

Safety assessments and measures of ADHD symptomatology will be collected prior to and during APZ therapy.

While receiving APZ treatment, patients will be seen at baseline, Week 1,2,3,4, and 6.

ELIGIBILITY:
Inclusion Criteria:

1. Outpatients ages 8-12 years (inclusive)
2. Currently meets DSM-IV (American Psychiatric Association, 1994) criteria for a primary diagnosis of ADHD (either predominantly inattentive type or combined type) based on the results of semi-structured diagnostic assessment (K-SADS-PL)(Kaufman et al., 1997) and based on the results of a clinical interview with a child and adolescent psychiatrist
3. Patients, who in the investigator's opinion, have substantial symptoms of ADHD for which pharmacotherapy is indicated
4. Has a guardian who has provided written informed consent to participate in this trial
5. Has provided written informed assent to participate in this study

Exclusion Criteria:

1. Patients who have a history of intolerance to APZ at a dose of 5 mg/day
2. Patients with a history of APZ allergy or hypersensitivity to APZ
3. Patients with an active or prior neurological/medical disorder for which treatment with APZ would be contraindicated (such as tardive dyskinesia or neuroleptic malignant syndrome)
4. Patients with clinical evidence of autistic disorder, Rett's syndrome or Asperger's syndrome
5. Patients with any bipolar spectrum disorder
6. Patients with any schizophrenia spectrum disorder
7. Patients with conduct disorder
8. Patients with post-traumatic stress disorder or generalized anxiety disorder
9. Patients with a substance abuse disorder
10. Females who are sexually active, pregnant or lactating
11. Patients with a suicide attempt requiring medical/psychiatric care within the past 6 months
12. Patient taking psychotropic agents within one week of baseline (3 days for psychostimulants, 2 weeks for fluoxetine)
13. Patients with evidence of mental retardation (I.Q. < 70) based on the results of the Peabody Picture Vocabulary Test- III (PPVT-III)(Dunn and Dunn, 1981)
14. Patients who have a general medical or neurological condition that could interfere with the interpretation of the clinical response to APZ treatment
15. Patients who are unable to swallow pills or capsules
16. Patients for whom the need for hospitalization during the course of the study appears likely

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 23 (Actual)
Dates: Start 2005-04; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Effectiveness and cognitive effects | 6 weeks
  To examine effectiveness and cognitive effects during open-label pilot

CONTACTS AND LOCATIONS:
Overall Officials: Robert L Findling, MD, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- University Hospitals Case Medical Center, Cleveland, Ohio, United States

REFERENCES:
- [Derived] Findling RL, Short EJ, Leskovec T, Townsend LD, Demeter CA, McNamara NK, Stansbrey RJ. Aripiprazole in children with attention-deficit/hyperactivity disorder. J Child Adolesc Psychopharmacol. 2008 Aug;18(4):347-54. doi: 10.1089/cap.2007.0124. PMID 18759644